CLINICAL TRIAL: NCT01733771
Title: Patient Reported Outcomes Following Complementary Medicine Treatments in Hospitalized Patients
Brief Title: The Effect of Complementary Medicine (CAM) Treatments on Common Symptoms in Hospitalized Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BNZ-0041-09
Record Dates: First submitted 2012-07-10; First posted 2012-11-27 (Estimated); Results first posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2019-07

CONDITIONS: Pain; Nausea; Anxiety
Keywords: complementary medicine; hospitalized
MeSH Terms: conditions — Pain; Nausea; Anxiety Disorders | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Reflexology (Experimental): Symptomatic hospitalized people randomized to reflexology on top of standard of care
  Interventions: Other: Reflexology
- Standard of care only (No Intervention): Symptomatic hospitalized people randomized to standard of care only
- Sham reflexology (Sham Comparator): Symptomatic hospitalized people randomized to sham reflexology on top of standard of care
  Interventions: Other: Sham reflexology

INTERVENTIONS:
Other: Reflexology — Reflexology intervention involved a 15-minute treatment in the induction room, provided by three reflexologists from the hospital staff. The reflexology protocol was developed through a Delphi method.
  Arms: Reflexology
Other: Sham reflexology — Sham reflexology intervention were given by two complementary medicine practitioners with knowledge in touch therapy (shiatsu) and included 15 minutes of gentle, nonspecific foot massage. Similarly to the true reflexology protocol, the protocol for this treatment was also determined in a consensus-reaching process among a group of four experienced reflexologists.
  Arms: Sham reflexology

SUMMARY:
This is a randomized, single blinded, interventional trial conducted in patients undergoing elective laparoscopic cholecystectomy, comparing the following three groups: Controls receiving standard-of-care (SoC) only (Group 1); intervention group receiving reflexology and SoC (Group 2); and a group receiving sham reflexology and SoC (Group 3). In all groups, level of preoperative anxiety was evaluated at entry and exit from the Holding Room Area (HRA). The evaluation was carried out using the Visual Analogue Scale for Anxiety (VAS-A) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years
2. Undergoing Laparoscopic Cholecysyectomy (LC)

Exclusion criteria:

1. Patients with a history of obstructive sleep apnea
2. Contraindication for benzodiazepines
3. Hemodynamic instability
4. Leg ulcers
5. Patients undergoing a LC together with another surgical procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2010-04; Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elad Schiff, Prof, Principal Investigator — Director, Internal Medicine B
Locations (1):
- Bnai Zion Medical Center, Haifa, Israel

REFERENCES:
- [Derived] Samuel A, Lital KB, Mostafa S, Ariel S, Yael G, Eran BA, Ibrahim M, Gideon S, Sagi G, Dan S, Elad S. Effectiveness of standard of care, vs. its combination with reflexology and sham reflexology on preoperative anxiety in patients undergoing elective laparoscopic cholecystectomy: a single-blinded randomized controlled trial. Front Med (Lausanne). 2025 Sep 12;12:1634575. doi: 10.3389/fmed.2025.1634575. eCollection 2025. PMID 41020221
- [Derived] Schiff E, Attias S, Matter I, Sroka G, Nae B, Arnon Z, Samuels N, Grinberg O, Ben-Arye E. Complementary and alternative medicine interventions for perioperative symptoms: A comparative effectiveness study. Complement Ther Med. 2019 Jun;44:51-55. doi: 10.1016/j.ctim.2019.03.003. Epub 2019 Mar 21. PMID 31126575

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Reflexology | Standard of Care Only | Sham Reflexology
Started | 101 | 100 | 99
Completed | 101 | 100 | 99
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reflexology | Standard of Care Only | Sham Reflexology | Total
Number analyzed (Participants) | 101 | 100 | 99 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (14.5) | 48.5 (15.3) | 49.9 (16.9) | 49.8 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 66 | 63 | 189
  Male | 41 | 34 | 36 | 111
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Number (percentage) of patients who received Anxiolytics: Diazepam or Oxazepam [Count of Participants; unit: Participants] | 23 | 25 | 24 | 72

OUTCOME MEASURES:

1. Primary Outcome: Perioperative Anxiety Expressed in Visual Analogue Scale for Anxiety (VAS-A) From 0 (Asymptomatic: no Anxiety) to 10 Extremely Symptomatic Anxiety
Description: Change of VAS-A between baseline and 4 hours post-treatment
Time Frame: Baseline and 4 hours post treatment: calculated as value at 4 hours post treatment minus value at baseline
Measure: Mean (Standard Deviation); unit: units on VAS-A scale
Arm/Group | Reflexology | Standard of Care Only | Sham Reflexology
Number analyzed (Participants) | 101 | 100 | 99
units on VAS-A scale | -2.83 (2.12) | 0.24 (1.06) | -1.99 (1.85)

ADVERSE EVENTS:
Time Frame: From baseline and until 1 year after recruitment
Arm/Group | Reflexology | Standard of Care Only | Sham Reflexology
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/100 | 0/99
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/100 | 0/99
Other Adverse Events (participants affected / at risk) | 0/101 | 0/100 | 0/99

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-15): https://cdn.clinicaltrials.gov/large-docs/71/NCT01733771/Prot_SAP_000.pdf